CLINICAL TRIAL: NCT02816606
Title: Radiological Follow-up of Alternative ACL Reconstruction Technique
Brief Title: Anterior Cruciate Ligament Radiology Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1610321; 16/SW/0080 (Other: South West Research Ethics Committee)
Record Dates: First submitted 2016-06-15; First posted 2016-06-28 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2016-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard Reconstruction Technique: ACL reconstruction using hamstring autograft Using 30-degree arthroscope Using rigid femoral tunnel reamer (Rigid Reamers)
- Alternative Reconstruction Group: ACL reconstruction using hamstring autograft Using 30-degree and 70-degree arthroscopes Using flexible femoral tunnel reamer (Flexible Reamers)
  Interventions: Procedure: Flexible reamers; Procedure: 70-degree arthroscope

INTERVENTIONS:
Procedure: Flexible reamers — These reamers allow creation of the femoral tunnel to be made in reduced knee flexion and potentially maximise tunnel length
  Groups: Alternative Reconstruction Group
Procedure: 70-degree arthroscope — Using this arthroscope (rather than the more traditional 30-degree) gives improved visualisation of the femoral and tibial footprints. This may translate into better positioning of the tunnel within these regions
  Groups: Alternative Reconstruction Group

SUMMARY:
Following recent advances in the understanding of successful anterior cruciate ligament (ACL) reconstruction, three important factors have been identified: femoral tunnel positioning, femoral tunnel aperture shape, and native remnant preservation. Accordingly, the researchers have adapted their technique to address these goals. This study is designed to assess the feasibility of evaluating these graft characteristics, on post-operative imaging, and the ability to show potential improvements with the researchers' technical changes. The study plans to use three-dimensional computer tomography (3D-CT) and magnetic resonance imaging (MRI) to assess these properties and the integration of the graft. In addition, the researchers will use their routine functional scores to monitor the patients' outcome. If successful, the research team hope to set-up a randomised control trial of this alternative technique versus conventional methods with assessment through the same imaging mediums and clinical follow-up.

DETAILED DESCRIPTION:
Rupture of the ACL has an incidence of 30 cases per 100,000 individuals in the UK. The number of reconstructions performed is increasing as more patients wish to maintain optimum knee function and stability, in older age-groups, than previously seen. The research centre (hospital) presently performs between 100 and 150 ACL reconstructions each year but, thus, this figure is likely to continue to rise.

The ACL performs a role in preventing anterior translation of the tibia on the femur, throughout the range of motion of the knee, but also provides rotational stability. Inadequate post-injury function, or failure, can result in continued feeling of instability (within the knee) and this may prevent return to employment as well as recreational activities. This is of particular importance to heavy manual workers and competitors in change-of-direction sports.

Reconstruction of the ACL most commonly involves the use of autologous hamstring or patellar tendon grafts that are implanted during an arthroscopic procedure. Rehabilitation, following reconstruction, is lengthy as the graft takes months to incorporate and over a year to regain mechanical properties. Therefore, these patients undergo a long period of functional rehabilitation, under the guidance of the physiotherapists, with repeated outpatient surgical follow-up to assess recovery and detect rare (but important) complications of surgery.

As understanding of the anatomy and biomechanics of the ACL has improved, the techniques used to perform this procedure have evolved accordingly. The goals of reconstructive surgery are to restore stability to the knee and allow the patient to return to employment and recreational activities. Research over the last 5 years has increasingly turned to defining the anatomy of this ligament and positioning the graft in an anatomical position. Bony landmarks have been identified for the position of the femoral footprint of the ACL - the intercondylar and bifurcate ridges - making positioning of the graft accurately possible. Appreciation of the importance of the remnant tissue - as an indication of previous attachment and as a conduit for revascularisation of the graft - and these bony landmarks for the tibial and femoral attachments, of the ligament, have led to changes in surgical philosophy and technique.

Of particular interest is the femoral tunnel. Successful ACL reconstruction has clearly been shown to be associated with femoral tunnel positioning so that the graft is centred in the original footprint and replicates the normal biomechanics of the knee. As there is a degree of variation between individuals, previous methods of positioning the graft relative to other structures (or using surrogate measurements) have been superseded by the need to identify these remaining anatomical landmarks. Therefore, operative technique has focussed on femoral footprint identification and centring the graft within this area.

Standard techniques, using a 30-degree arthroscope, provide limited views of both the femoral and tibial footprints. This is due to the orientation of these structures within the knee - parallel to the direction the arthroscope is introduced into the knee through the lateral portal. Remnant ACL tissue is removed, to improve visualisation and prevent impingement, as this was felt to be beneficial. As it is now recognised that remnant preservation is important, two conflicting challenges exist. The first is to improve visualisation whilst the second is to preserve the ACL stump as much as possible.

Attempts to improve the view obtained have led some surgeons to suggest introducing the arthroscope through a medial portal. However, this is not without additional problems such as instrument overcrowding and fluid leak from the knee. A 70-degree arthroscope increases the field of vision (particularly of structures parallel to the scope) without having to make additional portal sites. Therefore, the researchers have begun using this instrument within their team. Although, by improving the view, the researchers think this has improved positioning of the graft, it is difficult to assess either intra-operatively or on post-operative plain radiographs. 3D-CT is a validated and accurate tool for the assessment of femoral tunnel placement in the post-operative patient. Previous studies have been able to use this to measure the position of the tunnel, the tunnel aperture dimensions and the volume of the tunnel within the bone.

Visualisation can also be affected by the reamers used to create the tunnels for the graft. Traditional reamers are used over rigid wires. In order to introduce them into the knee, without causing damage to other structures, the knee must be maximally flexed. This leads to problems with the flow of the arthroscopy fluid (in a confined space) and may cloud of the operative field. This may be impossible to achieve in obese or well-muscled patients and the result is that some reaming takes place without a good view of positioning. A flexible reaming system can be used with the knee in a less flexed position further improving the view obtained. In addition, as the flexible guidewire (for the flexible reamers) enters the femoral wall more obliquely, the aperture created by the circular reamer is more oval in shape and length of the femoral tunnel may also be improved. This potentially means greater volume of graft within the femur and greater surface area for integration. The aperture shape, length and volume of this femoral tunnel can be further studied on the 3D-CT. This study of the femoral tunnel characteristics will be compared to both intra-operative assessments of position and size as, if there is good correlation, simpler techniques may be used in the future without the need for each patient to have a CT scan. A single CT study will be sufficient to make an assessment of these parameters for this study.

The research team have previously published a novel technique (using a 70-degree arthroscope) to achieve better visualisation of the footprints and give the surgeon a better chance of positioning the graft within the desired area (the native ACL footprint). Another group have published the combined technique of the 70-degree arthroscope and flexible reamers suggesting the advantages we anticipate in terms of tunnel characteristics. The researchers wish to formally evaluate the success of this alternative method against standard techniques.

The goal of ACL remnant preservation (and placement of the tunnels within this tissue) has been shown to result in increased revascularisation of the graft, increased cell-proliferation, and improved proprioception in the knee post-operatively. However, it has not been shown whether newer techniques (such as use of a 70-degree arthroscope and flexible reamers) impact on the ability of the surgeon to achieve this. Therefore, comparison of the healing rates and ligament appearances between those performed using this modified technique versus traditional methods is of interest. MRI is sensitive for the visualisation of soft-tissue structures. The researchers will, therefore, use this modality to evaluate the graft and remnant tissue. This will allow the research team to assess both position of the graft, within the remnant tissue, and integration of this graft over time. Other groups have been able to use MRI in this way to assess revascularisation of the graft and the maturation of graft material over time.

As the MRI will be used to assess graft integration, this will need to be repeated (throughout the follow-up period) to make serial measurements and quantify this progression.

If the researchers can show that it is feasible to replicate the previous successful use of MRI (as well as CT), and record a clear difference with the use of the flexible reamers and 70-degree arthroscope, they can lead on into a randomised control trial (RCT) of their technique versus standard methods. The researchers hope to demonstrate not only can CT and MRI be used to accurately measure graft position, tunnel shape and healing but also a difference between techniques in the main trial. As the standard techniques are used by other surgeons within the research team's department, this will provide the researchers with access to a comparative group. The team will be able to record results in both arms, which will provide information for conducting a full scale RCT. It will also allow for quantification of the changes the researchers can expect to be measuring, in an RCT, which will aid the power calculations required to guide recruitment numbers.

The required additional imaging can be timed with routine out-patient follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* All patients (Aged 18-50) undergoing ACL reconstruction in our unit

Exclusion Criteria:

* Age under 18 years
* Patient refusal following informed consent process
* Inability to undergo post-operative imaging (non-attendance, metal in body preventing MRI, pregnancy preventing CT)
* Different reconstruction technique chosen for clinical reasons.
* Revision procedures
* Previous surgery to the knee (or injury) that may affect the anatomy defined.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Anterior Cruciate Ligament rupture patients with clinical instability
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Anterior Cruciate Ligament Reconstruction Integrity | 12 months post-operative
  Assessed clinically and using MRI at 12 months post-operative

SECONDARY OUTCOMES:
Reamer size used for tibial and femoral tunnels | Intraoperative
  Reamer size in mm
Length of femoral tunnel | Intraoperative
  Length in mm - using arthroscopic ruler
Width of femoral tunnel | Intraoperative
  Width in mm - using arthroscopic ruler
Presence of Tibial Stump | Intraoperative
  Present or Absent
Dimensions of Femoral Tunnel | 3 months post-operative
  Measured on CT scan (in mm)
Aperture dimensions in femur | 3 months post-operative
  Measured on CT scan (in mm)
Position of femoral tunnel | 3 months post-operative
  Defined on 3-dimensional reconstruction of CT using grid-method
Revascularisation and healing of ACL graft | 3 months post-operative
  Assessed on MRI scan with signal comparison to posterior cruciate ligament
Revascularisation and healing of ACL graft | 12 months post-operative
  Assessed on MRI scan with signal comparison to posterior cruciate ligament

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Mandalia, MBBS, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon and Exeter Hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Dissemination in presentations at national meetings and publication in peer-reviewed journal

REFERENCES:
- [Background] Bucher TA, Naim S, Mandalia V. The use of the 70 degrees arthroscope for anatomic femoral and tibial tunnel placement and tunnel viewing in anterior cruciate ligament reconstruction. Arthrosc Tech. 2014 Jan 3;3(1):e79-81. doi: 10.1016/j.eats.2013.08.001. eCollection 2014 Feb. PMID 24749046
- [Background] Rasmussen JF, Lavery KP, Dhawan A. Anatomic anterior cruciate ligament reconstruction with a flexible reamer system and 70 degrees arthroscope. Arthrosc Tech. 2013 Aug 30;2(4):e319-22. doi: 10.1016/j.eats.2013.04.003. eCollection 2013. PMID 24400174
- [Result] Hosseini A, Lodhia P, Van de Velde SK, Asnis PD, Zarins B, Gill TJ, Li G. Tunnel position and graft orientation in failed anterior cruciate ligament reconstruction: a clinical and imaging analysis. Int Orthop. 2012 Apr;36(4):845-52. doi: 10.1007/s00264-011-1333-4. Epub 2011 Aug 9. PMID 21826407
- [Result] Tompkins M, Milewski MD, Carson EW, Brockmeier SF, Hamann JC, Hart JM, Miller MD. Femoral tunnel length in primary anterior cruciate ligament reconstruction using an accessory medial portal. Arthroscopy. 2013 Feb;29(2):238-43. doi: 10.1016/j.arthro.2012.08.019. Epub 2012 Dec 24. PMID 23270787
- [Result] Brown CH Jr, Spalding T, Robb C. Medial portal technique for single-bundle anatomical anterior cruciate ligament (ACL) reconstruction. Int Orthop. 2013 Feb;37(2):253-69. doi: 10.1007/s00264-012-1772-6. Epub 2013 Jan 20. PMID 23334708
- [Result] Gohil S, Annear PO, Breidahl W. Anterior cruciate ligament reconstruction using autologous double hamstrings: a comparison of standard versus minimal debridement techniques using MRI to assess revascularisation. A randomised prospective study with a one-year follow-up. J Bone Joint Surg Br. 2007 Sep;89(9):1165-71. doi: 10.1302/0301-620X.89B9.19339. PMID 17905952
- [Result] Ahn JH, Lee SH, Choi SH, Lim TK. Magnetic resonance imaging evaluation of anterior cruciate ligament reconstruction using quadrupled hamstring tendon autografts: comparison of remnant bundle preservation and standard technique. Am J Sports Med. 2010 Sep;38(9):1768-77. doi: 10.1177/0363546510368132. PMID 20805412
- [Result] Hong L, Li X, Zhang H, Liu X, Zhang J, Shen JW, Feng H. Anterior cruciate ligament reconstruction with remnant preservation: a prospective, randomized controlled study. Am J Sports Med. 2012 Dec;40(12):2747-55. doi: 10.1177/0363546512461481. Epub 2012 Oct 17. PMID 23075805
- [Result] Yang JH, Chang M, Kwak DS, Wang JH. Volume and contact surface area analysis of bony tunnels in single and double bundle anterior cruciate ligament reconstruction using autograft tendons: in vivo three-dimensional imaging analysis. Clin Orthop Surg. 2014 Sep;6(3):290-7. doi: 10.4055/cios.2014.6.3.290. Epub 2014 Aug 5. PMID 25177454
- [Result] Kim JG, Chang MH, Lim HC, Bae JH, Ahn JH, Wang JH. Computed tomography analysis of the femoral tunnel position and aperture shape of transportal and outside-in ACL reconstruction: do different anatomic reconstruction techniques create similar femoral tunnels? Am J Sports Med. 2013 Nov;41(11):2512-20. doi: 10.1177/0363546513500626. Epub 2013 Aug 27. PMID 23982402
- [Result] Forsythe B, Kopf S, Wong AK, Martins CA, Anderst W, Tashman S, Fu FH. The location of femoral and tibial tunnels in anatomic double-bundle anterior cruciate ligament reconstruction analyzed by three-dimensional computed tomography models. J Bone Joint Surg Am. 2010 Jun;92(6):1418-26. doi: 10.2106/JBJS.I.00654. PMID 20516317
- [Derived] Kosy JD, Walmsley K, Sharma AD, Gordon EA, Heddon SV, Anaspure R, Schranz PJ, Mandalia VI. A comparison of femoral tunnel placement in ACL reconstruction using a 70 degrees arthroscope through the anterolateral portal versus a 30 degrees arthroscope through the anteromedial portal: a pilot 3D-CT study. Knee Surg Relat Res. 2020 Apr 3;32(1):17. doi: 10.1186/s43019-020-00037-4. PMID 32660634